CLINICAL TRIAL: NCT05824143
Title: A Phase 1, Open-label, Fixed-Sequence Trial to Evaluate the Effect of Carbamazepine on the Single-Dose Pharmacokinetics of Darigabat in Healthy Adult Participants
Brief Title: Open-label Trial to Evaluate the Effect Carbamazepine on Darigabat Pharmacokinetics in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cerevel Therapeutics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CVL-865-HV-1003
Record Dates: First submitted 2023-03-24; First posted 2023-04-21 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Healthy Participants
MeSH Terms: interventions — Carbamazepine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Darigabat Followed by Darigabat + Carbamazepine (Experimental): Participants will receive darigabat tablet orally once on Day 1 of Treatment Period 1.
  Participants will receive carbamazepine tablets, titrated up to a steady-state dose, orally, twice daily (BID) from Day 1 to 17 along with the darigabat tablet orally once on Day 16 of Treatment Period 2.
  Interventions: Drug: Darigabat; Drug: Carbamazepine

INTERVENTIONS:
Drug: Darigabat — Oral tablet
  Other Names: CVL-865
Drug: Carbamazepine — Oral tablets

SUMMARY:
The primary purpose of the study is to evaluate the effect of increased metabolizing enzyme (cytochrome P450 [CYP] 3A4) due to carbamazepine, a strong CYP3A4 inducer, on the pharmacokinetics (PK) of darigabat in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Male and female (both women of childbearing and nonchildbearing potential) participants, ages 18-55 years, inclusive, at the time of signing the informed consent form (ICF).
* Sexually active women of childbearing potential must agree to be on a non-hormonal highly effective method of contraception with low user-dependency (eg, IUD or bilateral tubal ligation) from signing of informed consent throughout the duration of the trial until the last dose of darigabat and for an additional 33 days after the last dose of darigabat.

A male participant who is sexually active with a pregnant or a nonpregnant partner of childbearing potential must agree to use a condom during treatment and until the last dose of darigabat plus an additional 93 days. In addition, male participants should not donate sperm for a minimum of 93 days following last dose of darigabat.

* Healthy as determined by medical evaluation, including medical and psychiatric history, physical and neurological examinations, electrocardiogram (ECGs), vital sign measurements, and laboratory test results, as evaluated by the investigator.
* Body mass index of 18.5 to 35.0 kilograms per square meter (kg/m^2), inclusive, and total body weight ≥50 kilograms (kg) (110 pounds [lbs]) at Screening.
* Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the ICF.
* Ability, in the opinion of the investigator, to understand the nature of the trial and comply with protocol requirements, including the prescribed dosage regimens, scheduled visits, laboratory tests, and other trial procedures.

Exclusion Criteria:

* "Yes" responses for any of the following items on the Columbia-Suicide Severity Rating Scale (C-SSRS) (within the individual's lifetime):

  * Suicidal Ideation Item 3 (Active Suicidal Ideation with Any Methods [Not Plan] without Intent to Act)
  * Suicidal Ideation Item 4 (Active Suicidal Ideation with Some Intent to Act, without Specific Plan)
  * Suicidal Ideation Item 5 (Active Suicidal Ideation with Specific Plan and Intent)
  * Any of the Suicidal Behavior items (Actual Attempt, Interrupted Attempt, Aborted Attempt, Preparatory Acts or Behavior) "Yes" responses for any of the following items on the C-SSRS (within past 12 months):
  * Suicidal Ideation Item 1 (Wish to be Dead)
  * Suicidal Ideation Item 2 (Non-Specific Active Suicidal Thoughts) Serious risk of suicide in the opinion of the investigator is also exclusionary.
* Any condition or surgery that could possibly affect drug absorption, including, but not limited to, bowel resections, bariatric weight loss surgery/procedures, gastrectomy, and cholecystectomy.
* Known allergy or hypersensitivity to the investigational medicinal product (IMP), including carbamazepine, closely related compounds, or any of their specified ingredients.
* Participants positive for human leukocyte antigen (HLA)-B 1502 or HLA-A 3101.
* Use of prohibited medication prior to randomization (5 half-lives) or likely to require prohibited concomitant therapy during the trial. CYP3A4 inhibitors and inducers are prohibited from 30 days prior to signing of the ICF through the end of the trial. Vaccinations or boosters within 7 days of planned dosing or while on trial are prohibited.
* Recent monoamine oxidase (MAO)-I use (in the last 28 days), as it increases the risk for hypersensitivity and bone marrow suppression from carbamazepine.
* Prior carbamazepine use that was discontinued for tolerability or adverse events, including a clinically significant decrease in platelets, white blood cells, or hemoglobin.
* Any of the following clinical laboratory test results at the Screening Visit or Check-in (Day -1), which can be confirmed by a single repeat measurement:

  * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > upper limit of normal (ULN)
  * Total bilirubin >1.5 × ULN. If Gilbert's syndrome is suspected, total bilirubin > ULN is acceptable if the conjugated or direct bilirubin fraction is <20% of total bilirubin, and eligibility is confirmed following discussion with the medical monitor.
* Any of the following clinical laboratory test results at the Screening Visit or Check-in (Day -1), which can be confirmed by a single repeat measurement:

  * Platelets, white blood cell count, absolute neutrophil count, or hemoglobin < lower limit of normal (LLN)
  * Serum sodium < LLN

Note: Other protocol-defined exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2023-04-17 (Actual); Primary Completion 2023-07-07 (Actual); Study Completion 2023-07-07 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of Darigabat | Treatment Period 1: 15 minutes pre-dose on Day 1 and up to 48 hours post dose; Treatment Period 2: 15 minutes pre-dose on Day 16 and up to 48 hours post dose
  PK of darigabat will be analyzed both in the presence and absence of carbamazepine.
Area Under the Plasma Concentration-time Curve up to the Last Specified Sampling Time (AUC0-t) of Darigabat | Treatment Period 1: 15 minutes pre-dose on Day 1 and up to 48 hours post dose; Treatment Period 2: 15 minutes pre-dose on Day 16 and up to 48 hours post dose
  PK of darigabat will be analyzed both in the presence and absence of carbamazepine.
Area Under the Plasma Concentration-time Curve From Time 0 to Infinity (AUCinf) of Darigabat | Treatment Period 1: 15 minutes pre-dose on Day 1 and up to 48 hours post dose; Treatment Period 2: 15 minutes pre-dose on Day 16 and up to 48 hours post dose
  PK of darigabat will be analyzed both in the presence and absence of carbamazepine.

SECONDARY OUTCOMES:
Number of Participants With Treatment-emergent Adverse Events (TEAEs) | Up to Day 52
Number of Participants with Clinically Significant Changes in Electrocardiogram (ECG) Values | Up to Day 21
Number of Participants With Clinically Significant Changes in Vital Sign Values | Up to Day 21
Number of Participants With Clinically Significant Changes in Clinical Laboratory Assessments | Up to Day 21
Number of Participants With Clinically Significant Changes in Physical and Neurological Examination Results | Up to Day 21
Changes in Suicidality Assessed Using the Columbia Suicide Severity Rating Scale (C-SSRS) | Up to Day 21
  The C-SSRS includes 'yes' or 'no' responses for assessment of suicidal ideation and behavior as well as numeric ratings for severity of ideation, if present (from 1 to 5, with 5 being the most severe). Greater lethality or potential lethality of suicidal behaviors (endorsed on the behavior subscale) indicates increased risk.

CONTACTS AND LOCATIONS:
Locations (1):
- Orlando, Florida, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No